CLINICAL TRIAL: NCT02151682
Title: An Open-label Trial, Enrolling Subjects Aged 6 Years to Less Than 18 Years Suffering From Pain Requiring Prolonged Release Opioid Treatment, to Evaluate the Safety and Efficacy of Tapentadol PR Versus Morphine PR, Followed by an Open-label Extension
Brief Title: A Study to Look at Tapentadol Tablets in Children and Adolescents in Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KF5503-66; 2012-004360-22 (EudraCT Number); U1111-1154-4572 (Other: WHO)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Pain
Keywords: chronic pain; opioid
MeSH Terms: conditions — Pain; Chronic Pain | interventions — Tapentadol

STUDY DESIGN:
Intervention Model Description: There were 2 arms in Part 1: Randomization was carried out in blocks and in a 2:1 ratio (tapentadol PR to morphine PR). Participants were stratified using interactive response technology: by age group (6 years to less than 12 years and 12 years to less than 18 years, at the second visit [Allocation Visit]) so that at least 25% of participants were in the younger age group, and by underlying pain condition (cancer/non-cancer-related pain).
  There were 4 arms in Part 2: The investigators/participants decided if participants from Part 1 switched to or continued on tapentadol PR (tapentadol arm) or if they received no treatment/standard of care treatment if needed (2 direct observation arms following treatment in Part 1 and 1 observation arm after initial treatment with tapentadol in Part 2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Morphine prolonged-release (Part 1) (Active Comparator): 10 milligram (mg) or 30 mg tablets were taken orally twice daily. Starting doses varied from 10 to 40 mg morphine PR twice daily depending on participant's weight; if necessary, doses were gradually increased up to a maximum dose defined per weight group.
  The highest dose defined for participants weighing 55 kg and more was 200 mg per day.
  Interventions: Drug: Morphine prolonged release
- Tapentadol prolonged-release (Part 1) (Experimental): 25 mg or 100 mg tablets were taken orally twice daily. Starting doses varied from 25 to 100 mg tapentadol PR twice daily depending on participant's weight. If necessary, doses were gradually increased up to a maximum dose defined per weight group.
  The highest dose defined for participants weighing 55 kg and more was 500 mg per day.
  Interventions: Drug: Tapentadol prolonged release
- Tapentadol in Part 2 after Tapentadol or Morphine in Part 1 (Experimental): Participants on tapentadol PR in Part 1 of the study continued on the current dose of tapentadol PR in Part 2 and if necessary could modify their tapentadol PR dosage. Participants who were randomized to morphine PR in Part 1 of the study were rotated to tapentadol PR in Part 2 with 70 percent of their current morphine equivalent dose or lower. The dosage could be increased gradually up to approximately 4.5 mg/kg body weight tapentadol PR twice daily.
  Interventions: Drug: Tapentadol prolonged release
- Observation Period after Tapentadol in Part 1 (No Intervention): Participants who completed tapentadol PR in Part 1 of the study or discontinued tapentadol treatment early in Part 1 could continue directly in the observation period in Part 2 for up to 12 months (with standard-of-care treatment if needed).
- Observation Period after Morphine in Part 1 (No Intervention): Participants who completed morphine PR treatment in Part 1 of the study or discontinued early from morphine treatment in Part 1 could continue directly in the observation period in Part 2 (with standard-of-care treatment if needed).
- Observation Period after Tapentadol in Part 2 (No Intervention): Participants who completed tapentadol PR or morphine PR treatment in Part 1 of the study could enter the Observation Period for up to 12 months (with standard-of-care treatment if needed) after they had discontinued from tapentadol PR treatment in Part 2.

INTERVENTIONS:
Drug: Tapentadol prolonged release
  Other Names: Palexia®; Nucynta®; Yantil®
  Arms: Tapentadol in Part 2 after Tapentadol or Morphine in Part 1; Tapentadol prolonged-release (Part 1)
Drug: Morphine prolonged release
  Arms: Morphine prolonged-release (Part 1)

SUMMARY:
Tapentadol has already been studied in adults. This study is needed to find out if tapentadol works and is safe to use in children and adolescents with long-term pain.

DETAILED DESCRIPTION:
During the first 2 weeks of the study (Part 1), participants were given either tapentadol or morphine prolonged-release (PR) tablets. Assignment was done randomly (like tossing a coin). The participant and the caregiver knew which medication the child was taking. The primary endpoint was based on data collected in Part 1 of this study.

If eligible and willing, participants from Part 1 could enter a 12 month follow-up period (Part 2). In Part 2 of this study, participants were either treated with tapentadol PR tablets or entered observations arms where they were not treated at all or with standard of care.

ELIGIBILITY:
Inclusion Criteria:

Part 1 - Randomized to open-label, active comparator controlled treatment

Participants were eligible for the study at enrollment if all the following applied:

* Informed consent (if applicable assent) obtained.
* Male or female participant at least 6 years of age at the Enrollment Visit and less than 18 years of age on Day 14.
* Participant has an underlying long-term pain condition (e.g., cancer, chronic disease, planned or performed surgery) that is, according to the judgment of the investigator, expected to require a twice-daily prolonged release opioid treatment until at least the end of the 14-day Treatment Period.
* Participant can swallow tablets of appropriate size.
* Participant is able to participate in the study as planned and willing to comply with the requirements of the protocol including refraining from drinking beverages containing alcohol and recreational intake of drugs while on study medication.

Participants had to satisfy the following criteria before allocation to treatment:

* Less than 18 years of age.
* No opioid intake or last calculated morphine equivalent dose of less than 3.5 mg/kg per day.
* Participant has a body weight of at least 17.5 kg.
* If a female of childbearing potential (post menarchal and not surgically incapable of childbearing) and sexually active, must practice an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double barrier method, contraceptive patch) before allocation to study medication until the end of intake of study medication.
* If a female and post menarchal or older than 12 years, has a negative urine pregnancy test on the day before or on the day of allocation to study medication.

Part 2

Inclusion criteria for the Tapentadol Open-label extension period:

* Participant has completed the 14-day Treatment Period.
* Participant is still in need of prolonged release opioid treatment.
* Participant does not meet any of the compulsory discontinuation criteria.

Exclusion Criteria:

Participants were not eligible for the study if any of the following applied.

The following was checked at enrollment:

* Has been previously enrolled in this study or a previous study with tapentadol.
* Has a clinically relevant history of hypersensitivity, allergy, or contraindication to morphine or tapentadol or any ingredient, including galactose intolerance (see investigator's brochure for tapentadol prolonged-release [PR] and summary of product characteristics for morphine PR), or naloxone.
* History or current condition of any one of the following:

  * Seizure disorder or epilepsy.
  * Serotonin syndrome.
  * Traumatic or hypoxic brain injury, brain contusion, stroke, transient ischemic attack, intracranial hematoma, posttraumatic amnesia, brain neoplasm, or episode(s) of more than 24 hours duration of unconsciousness.
* History or current condition of any one of the following:

  * Moderate to severe renal or hepatic impairment.
  * Abnormal pulmonary function or clinically relevant respiratory disease (e.g., acute or severe bronchial asthma, hypercapnia)
  * Complex regional pain syndrome.
  * A pain indication with a strong psycho-somatic component that, in the judgment of the investigator, is unlikely to respond to opioids.
* History of alcohol or drug abuse in the investigator's judgment, based on history and physical examination. Drugs of abuse detected in urine screen unless explained by allowed concomitant medication
* Participant has:

  * A clinically relevant abnormal electrocardiogram.
  * Signs of pre-excitation syndrome.
  * Brugada's syndrome.
  * QT or corrected QT (QTcF, Fridericia) interval greater than 470 ms.
* Any surgery scheduled during the first 14 days of the study that is expected to require post-surgical intensive care unit (ICU) treatment, or that requires post-surgical parenteral pain-treatment, or may, affect the safety of the participant.
* Participant is not able to understand and comply with the protocol as appropriate for the age of the participant or participant is cognitively impaired in the investigator's judgment such that they cannot comply with the protocol.
* Participant, parent or the legal representative is an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, or family member of the employees or the investigator.

The following was checked at the enrollment and the allocation visits:

* Has a concomitant disease or disorder (e.g., endocrine, metabolic, neurological, psychiatric, infection) that in the opinion of the investigator may affect or compromise participant safety during the study participation.
* Pancreatic/biliary tract disease (e.g., pancreatitis) or paralytic ileus.
* Intake of forbidden concomitant medication/use of forbidden therapies (see synopsis section Concomitant medications/therapies).
* Female participant is breastfeeding a child.

The following was checked at the allocation to treatment visit:

* Has received a drug or used a medical device not approved for human use within 30 days prior to visit.
* Based on data from the local laboratory, one or more of:

  * Total serum bilirubin greater than 2.0 mg/dL.
  * Serum albumin less than 2.8 g/dL.
  * Aspartate transaminase or alanine transaminase greater than 5 times upper limit of normal.
* Based on data from the local laboratory, creatinine clearance less than 30 mL/min per 1.73 m2 (calculated according to a formula that is appropriate for the respective age group).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Trials, Study Director — Grünenthal GmbH
Locations (23):
- BE001, Leuven, Belgium
- Bulgaria (4):
  - BG005, Pleven
  - BG004, Plovdiv
  - BG001, Sofia
  - BG006, Sofia
- Chile (2):
  - CL004, Santiago
  - CL001, Valparaíso
- France (7):
  - FR008, Amiens
  - FR004, Brest
  - FR002, Lille
  - FR006, Lyon
  - FR005, Nice
  - FR001, Vandœuvre-lès-Nancy
  - FR003, Villejuif
- DE001, Homburg, Germany
- HU001, Budapest, Hungary
- IT003, Turin, Italy
- Portugal (2):
  - PT001, Braga
  - PT002, Porto
- ES003, Valladolid, Spain
- United Kingdom (3):
  - GB005, Leeds
  - GB003, Manchester
  - GB006, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Web Site (see URL below for details)
Supporting Information: Study Protocol, SAP, CSR
URL: http://www.grunenthal.com/r-d-vision-mission/clinical-trials/data-sharing-clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled for Part 1 on 29 April 2015.
Pre-assignment Details: 73 participants signed an informed consent form (assented). 1 participant withdrew consent and 2 did not meet in-/exclusion criteria. 70 participants were allocated to investigational medicinal product (IMP). 1 of the allocated participants was not treated, resulting in 69 participants who were dosed in Part 1.
Groups:
- Tapentadol in Part 2 After Tapentadol or Morphine in Part 1: 26 Participants on tapentadol PR in Part 1 continued on the current dose of tapentadol PR in Part 2 and if necessary could modify their tapentadol PR dosage. 10 Participants on morphine PR in Part 1 were rotated to tapentadol PR in Part 2 with 70 percent of their current morphine equivalent dose or lower. The dosage could be increased gradually up to approximately 4.5 mg/kg body weight tapentadol PR twice daily.
  Treatment with tapentadol was up to 12 months in Part 2.
- Observation Period After Tapentadol in Part 1: 14 Participants who completed tapentadol PR in Part 1 of the study and 4 of 5 participants who discontinued tapentadol treatment early in Part 1 continued directly in the observation period in Part 2 for up to 12 months (with standard-of-care treatment if needed).
  One subject who withdrew consent in Part 1 did not enter the observation period.
- Observation Period After Morphine in Part 1: 12 Participants who completed morphine PR treatment in Part 1 of the study and 2 participants who discontinued early from morphine treatment in Part 1 continued directly in the observation period in Part 2 (with standard-of-care treatment if needed).
- Observation Period After Tapentadol in Part 2: 19 Participants who completed tapentadol treatment in Part 1 and discontinued from tapentadol treatment in Part 2 and 7 participants who completed morphine treatment in Part 1 and discontinued from tapentadol in Part 2 entered the Observation Period for up to 12 months (with standard-of-care treatment if needed).
Period: Part 1: 14 Days Morphine or Tapentadol
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1) | Tapentadol in Part 2 After Tapentadol or Morphine in Part 1 | Observation Period After Tapentadol in Part 1 | Observation Period After Morphine in Part 1 | Observation Period After Tapentadol in Part 2
Started | 24 | 45 | 0 (Group not defined for Part 1.) | 0 (Group not defined for Part 1.) | 0 (Group not defined for Part 1.) | 0 (Group not defined for Part 1.)
Completed | 22 (14-Day treatment and final post-treatment visit completed or tapentadol treatment in Part 2 entered.) | 40 (14-Day treatment and final post-treatment visit completed or tapentadol treatment in Part 2 entered.) | 0 | 0 | 0 | 0
Not Completed | 2 | 5 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Technical problems | 0 | 1 | 0 | 0 | 0 | 0
Not completed — No need for opioid | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Missing | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Tapent. Extension or Observation
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1) | Tapentadol in Part 2 After Tapentadol or Morphine in Part 1 | Observation Period After Tapentadol in Part 1 | Observation Period After Morphine in Part 1 | Observation Period After Tapentadol in Part 2
Started | 0 (Group not defined for Part 2.) | 0 (Group not defined for Part 2.) | 36 (26 Completers on tapentadol PR and 10 completers on morphine PR from Part 1.) | 18 (14 Completers and 4 of 5 non-completers on tapentadol in Part 1.) | 14 (12 Completers and 2 non-completers from morphine treatment in Part 1.) | 0
Completed | 0 | 0 | 8 (12 Month of tapentadol treatment completed and final visit of Part 2 performed.) | 14 | 14 | 0
Not Completed | 0 | 0 | 28 | 4 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — No need for opioid | 0 | 0 | 13 | 0 | 0 | 0
Not completed — Missing | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Various other | 0 | 0 | 6 | 0 | 0 | 0
Not completed — Final post-treatment visit not performed | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 2: Observ. Aft. Tapent. Extension
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1) | Tapentadol in Part 2 After Tapentadol or Morphine in Part 1 | Observation Period After Tapentadol in Part 1 | Observation Period After Morphine in Part 1 | Observation Period After Tapentadol in Part 2
Started | 0 (Group not defined for Part 2.) | 0 (Group not defined for Part 2.) | 0 (Not applicable for this period.) | 0 (Not applicable for this period.) | 0 (Not applicable for this period.) | 26 (19 tapentadol and 7 morphine completers (Part 1) who discontinued from tapentadol treatm. in Part 2.)
Completed | 0 | 0 | 0 | 0 | 0 | 19
Not Completed | 0 | 0 | 0 | 0 | 0 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Missing | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Various other | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Set
Groups:
- Morphine Prolonged-release (Part 1): The treatment group comprised 7 participants aged 6 years to less than 12 years and 17 participants aged 12 years to less than 18 years.
  Starting doses varied from 10 to 40 milligrams (mg) morphine PR twice daily depending on participant's weight; if necessary, doses were gradually increased up to a maximum dose defined per weight group.
  The highest dose defined for participants weighing 55 kg and more was 200 mg per day.
- Tapentadol Prolonged-release (Part 1): The treatment group comprised 12 participants aged 6 years to less than 12 years and 33 participants aged 12 years to less than 18 years.
  Starting doses varied from 25 to 100 mg tapentadol PR twice daily depending on participant's weight. If necessary, doses were gradually increased up to a maximum dose defined per weight group.
  The highest dose defined for participants weighing 55 kg and more was 500 mg per day.
- Total: Total of all reporting groups
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1) | Total
Number analyzed (Participants) | 24 | 45 | 69
Age, Continuous [Mean (Standard Deviation); unit: years]
  All participants | 13.2 (2.8) | 13.2 (2.8) | 13.2 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 22 | 32
  Male | 14 | 23 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 20 | 36 | 56
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 24 | 44 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Age, customized [Count of Participants; unit: Participants]
  6 years to less than 12 years | 7 | 12 | 19
  12 years to less than 18 years | 17 | 33 | 50
Height [Mean (Standard Deviation); unit: centimeters] — Population: Height is presented by age group.
  centimeters
    6 years to less than 12 years: number analyzed (Participants) | 7 | 12 | 19
    6 years to less than 12 years | 138.9 (13.4) | 136.0 (12.5) | 137.1 (12.5)
    12 years to less than 18 years: number analyzed (Participants) | 17 | 33 | 50
    12 years to less than 18 years | 165.8 (11.2) | 162.9 (11.3) | 163.9 (11.2)
Weight [Mean (Standard Deviation); unit: kilograms] — Population: Weight is presented by age group.
  kilograms
    6 years to less than 12 years: number analyzed (Participants) | 7 | 12 | 19
    6 years to less than 12 years | 34.17 (14.08) | 32.37 (11.39) | 33.03 (12.09)
    12 years to less than 18 years: number analyzed (Participants) | 17 | 33 | 50
    12 years to less than 18 years | 56.69 (9.52) | 56.35 (13.92) | 56.47 (12.50)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Body Mass Index is presented by age group.
  kg/m^2
    6 years to less than 12 years: number analyzed (Participants) | 7 | 12 | 19
    6 years to less than 12 years | 17.28 (5.69) | 17.08 (3.38) | 17.16 (4.22)
    12 years to less than 18 years: number analyzed (Participants) | 17 | 33 | 50
    12 years to less than 18 years | 20.59 (2.98) | 21.15 (4.66) | 20.96 (4.14)
Pain cause [Count of Participants; unit: Participants] — Population: As a parameter of special interest, pain cause (cancer-related pain, non-cancer-related pain) was presented by age group.
  Participants
    Cancer-related pain: number analyzed (Participants) | 5 | 9 | 14
    Cancer-related pain: 6 years to less than 12 years | 1 | 0 | 1
    Cancer-related pain: 12 years to less than 18 years | 4 | 9 | 13
    Non-cancer-related pain: number analyzed (Participants) | 19 | 36 | 55
    Non-cancer-related pain: 6 years to less than 12 years | 6 | 12 | 18
    Non-cancer-related pain: 12 years to less than 18 years | 13 | 24 | 37
Type of pain [Count of Participants; unit: Participants]
  Neuropathic | 4 | 9 | 13
  Nociceptive/somatic | 13 | 28 | 41
  Nociceptive/visceral | 0 | 0 | 0
  Neuropathic and nociceptive/somatic | 6 | 6 | 12
  Neuropathic and nociceptive/visceral | 0 | 0 | 0
  Nociceptive/somatic and nociceptive/visceral | 1 | 1 | 2
  All of the pain types | 0 | 1 | 1
Pain intensity (FPS-R) [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was assessed on a revised Faces Pain Scale (FPS-R). The FPS-R is a validated self-reported 6 point scale with 0 representing "no pain" and 10 representing "very much pain". Facial representations are used to indicate how much the pain hurts. Population: FPS-R data at baseline were available for 32 participants on tapentadol PR and for 19 participants on morphine PR (51 of 69 participants overall).
  units on a scale
    6 years to less than 12 years: number analyzed (Participants) | 6 | 10 | 16
    6 years to less than 12 years | 6.7 (2.1) | 5.8 (3.6) | 6.1 (3.1)
    12 years to less than 18 years: number analyzed (Participants) | 13 | 22 | 35
    12 years to less than 18 years | 3.1 (2.7) | 4.0 (3.1) | 3.7 (2.9)
Pain intensity (VAS) [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to indicate the current level of pain intensity at the time of assessment on a validated vertical Visual Analog Scale (VAS). It was scored such that a score of 0 was equivalent to "no pain" and a score of 100 was equivalent to "pain as bad as it could be". Population: VAS data at baseline were available for 32 participants on tapentadol PR and for 19 participants on morphine PR (51 of 69 participants overall).
  units on a scale
    6 years to less than 12 years: number analyzed (Participants) | 6 | 10 | 16
    6 years to less than 12 years | 75.3 (14.6) | 59.1 (32.8) | 65.2 (28.0)
    12 years to less than 18 years: number analyzed (Participants) | 13 | 22 | 35
    12 years to less than 18 years | 39.5 (32.4) | 42.7 (31.6) | 41.5 (31.5)
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 0 | 1 | 1
  Italy | 0 | 3 | 3
  Portugal | 4 | 3 | 7
  Spain | 1 | 1 | 2
  United Kingdom | 1 | 7 | 8
  Chile | 3 | 4 | 7
  France | 5 | 9 | 14
  Germany | 4 | 5 | 9
  Belgium | 0 | 1 | 1
  Bulgaria | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified as Responder (Part 1)
Description: The proportion of participants classified as responders was assessed and compared between the treatment groups.
  A participant was defined as responder if both of the following criteria were met:
  * Completion of the 14-day Treatment Period (Part 1).
  * One of the following calculated from the scheduled pain assessments ("pain right now") documented during the last 3 days of the Treatment Period:
    * Average pain less than 50 on a visual analog scale (VAS, range 0 [no pain] to 100 [pain as bad as it could be]) for participants aged 12 years to less than 18 years; or less than 5 on the Faces Pain Scale-revised (FPS-R, range 0 [no pain] and 10 [very much pain]) for participants aged 6 years to less than 12 years.
    * Average reduction from baseline of pain greater than or equal to 20 on a VAS for participants aged 12 years to less than 18 years; or greater than or equal to 2 on the FPS-R for participants aged 6 years to less than 12 years.
Time Frame: From Day 1 up to Day 14 (End of Part 1)
Population: Full Analysis Set; missing pain assessments (last 3 days) were imputed using multiple imputation.
Measure: Count of Participants; unit: Participants
Groups:
- Tapentadol Prolonged-release (Part 1): The treatment group comprised 12 participants aged 6 years to less than 12 years and 33 participants aged 12 years to less than 18 years. Participants starting doses varied from 25 to 100 mg tapentadol PR twice daily depending on participant's weight. If necessary, doses were gradually increased up to a maximum dose defined per weight group.
  The highest dose defined for participants weighing 55 kg and more was 500 mg per day.
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1)
Number analyzed (Participants) | 24 | 45
Participants | 19 | 32
Statistical Analysis 1: Comparison: Morphine Prolonged-release (Part 1) vs Tapentadol Prolonged-release (Part 1); Test type: Non-Inferiority — A logistic regression model was fitted to the response using baseline pain, age group, treatment, and underlying pain condition as explanatory variables, followed by a Farrington-Manning test for non-inferiority, based on Full Analysis Set; p = 0.0790, Farrington-Manning test — The p-value is based on Farrington-Manning variance estimator using a pre-specified non-inferiority margin of -0.2. A 1-sided alpha of 0.1 was used. A p-value <0.1 represents non-inferiority; Non-inferiority of tapentadol prolonged-release versus morphine prolonged-release has been demonstrated; Risk Difference (RD) = -0.06, 80% CI 2-sided [-0.19 to 0.06] — A confidence interval for the risk difference (RD) completely above the pre-specified non-inferiority margin of -0.2 represents non-inferiority of tapentadol prolonged-release versus morphine prolonged-release

2. Secondary Outcome: Extent of Constipation (Part 1)
Description: Constipation was assessed using the modified constipation assessment scale (mCAS). This is an 8-item questionnaire where the observer has scored constipation on a nominal scale (no Problem [score 0], some problem [score 1] or severe Problem [score 2]). The response to an item could also be scored as "unable to assess".
  The Total Score can vary from 0-16; the higher the Total Score the higher the extent of constipation. A positive change from Day 1 to Day 14 indicates a worsening, a negative change an improvement.
Time Frame: From Day 1 to Day 14 (End of Part 1)
Population: Safety Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1)
Number analyzed (Participants) | 24 | 45
score on a scale
  Day 1: number analyzed (Participants) | 23 | 40
  Day 1 | 2.7 (3.0) | 1.5 (1.4)
  Day 14: number analyzed (Participants) | 24 | 41
  Day 14 | 2.7 (2.4) | 1.8 (2.0)
  Change from Day 1: number analyzed (Participants) | 23 | 39
  Change from Day 1 | -0.1 (1.6) | 0.4 (2.4)

3. Secondary Outcome: Tolerability Over the Complete Trial Period
Description: Tolerability was assessed by the number of participants with exactly 1 to more than 5 treatment emergent adverse events (TEAE) by treatment group during the different trial periods, on a participant level.
  In addition, tolerability was assessed by the number of participants with TEAEs which were considered by the investigator to be at least possibly related to the treatment the participant received.
Time Frame: Part 1: Day 1 (Start of Part 1) to Day 14; Part 2: Day 15 to Day 379 (End of Part 2)
Population: Safety Set
Measure: Number; unit: participants
Groups:
- Tapentadol Prolonged-release (Part 2): 36 Participants who completed Part 1 of the trial (26 on tapentadol PR and 10 participants on morphine PR) continued treatment or switched to treatment with tapentadol PR for up to 12 months in Part 2.
  Participants on tapentadol PR in Part 1 continued on the current dose of tapentadol PR in Part 2 and if necessary could modify their tapentadol PR dosage. Participants on morphine PR in Part 1 were rotated to tapentadol PR in Part 2 with 70 percent of their current morphine equivalent dose or lower. The dosage could be increased gradually up to approximately 4.5 mg/kg body weight tapentadol PR twice daily.
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 2)
Number analyzed (Participants) | 24 | 45 | 36
participants
  Participants without any TEAE | 12 | 19 | 6
  Participants with at least 1 TEAE | 12 | 26 | 30
  Participants with exactly 1 TEAE | 1 | 7 | 5
  Participants with exactly 2 TEAEs | 2 | 5 | 2
  Participants with exactly 3 TEAEs | 2 | 4 | 2
  Participants with exactly 4 TEAEs | 2 | 1 | 4
  Participants with exactly 5 TEAEs | 1 | 3 | 3
  Participants with more than 5 TEAEs | 4 | 6 | 14
  Participants with related TEAEs | 6 | 12 | 13

4. Other Pre Specified Outcome: Change in Pain Intensity in the Open-label, Active-controlled Treatment Period (Part 1)
Description: Pain intensity was assessed by scoring "Pain right now" twice daily up to Day 14 by every participant using the Visual Analog Scale (VAS) as well as the Faces Pain Scale-Revised (FPS-R) in an electronic diary. Pain intensity was first documented using the VAS and directly thereafter the FPS-R. If required, pain intensity diary entry could be assisted by the legal guardian or a health care provider.
  The VAS is scored from 0, equivalent to "no pain", to 100, equivalent to "pain as bad as it could be".
  The FPS-R is a validated self-reported 6-point scale with 0 representing "no pain" and 10 representing "very much pain". Facial representations were used to indicate how much the pain hurts.
  The "pain right now" scores at baseline (last evaluation before starting IMP) and the mean of last 6 assessments collected up to the time point of last IMP intake in Part 1 (i.e., Day 14 or the day of early discontinuation) were used for the calculation of the change in pain intensity from baseline.
Time Frame: From Baseline up to Day 14 (End of Part 1) or early discontinuation
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1)
Number analyzed (Participants) | 24 | 45
units on a scale
  Pain intensity change from Baseline (FPS-R): number analyzed (Participants) | 17 | 29
  Pain intensity change from Baseline (FPS-R) | -2.0 (3.5) | -1.9 (3.4)
  Pain intensity change from Baseline (VAS): number analyzed (Participants) | 17 | 29
  Pain intensity change from Baseline (VAS) | -23.4 (36.9) | -18.8 (33.5)

5. Other Pre Specified Outcome: Change in Pain Intensity in the Tapentadol Open-label Extension Period (Part 2)
Description: Pain intensity was assessed by scoring "Pain right now" using the Visual Analog Scale (VAS) as well as the Faces Pain Scale-Revised (FPS-R) at each visit. The pain intensity was first documented using the VAS and directly thereafter the FPS-R. If required, pain intensity assessments could be assisted by the legal guardian or a health care provider.
  The VAS is scored from 0, equivalent to "no pain", to 100, equivalent to "pain as bad as it could be". The FPS-R is a validated self-reported 6-point scale with 0 representing "no pain" and 10 representing "very much pain". Facial representations were used to indicate how much the pain hurts.
  The "pain right now" score at the tapentadol baseline (last evaluation before or at Day 15) and at the last assessment for those subjects who completed the 12 months treatment of Part 2 were used for the calculation of the change in pain intensity from the tapentadol baseline.
Time Frame: From Day 15 to Day 379 (End of Part 2)
Population: Full Analysis Set; data from 9 subjects who completed the visit 12 months after start of Part 2 were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol Prolonged-release (Part 2)
Number analyzed (Participants) | 9
units on a scale
  Pain intensity change (FPR-S) from Day 15 | 0 (2.8)
  Pain intensity change (VAS) from Day 15 | -11.7 (29.0)

6. Other Pre Specified Outcome: Use of Rescue Medication in the Open-Label, Active-controlled Treatment Period (Part 1)
Description: Due to an overall low intake of rescue medication, it was not appropriate to present the number of doses of oral morphine solution used at different dose levels of investigational medicinal product (IMP) but the average daily dose (milligrams per kilogram body weight) for the treatment period and a modified average daily dose. Average daily dose and modified average daily dose were both calculated based on drug accountability.
  For the modified average daily doses, implausible values were excluded from the analysis, i.e., the amount of rescue medication that was lost due to a broken bottle was excluded from the analysis and negative amounts of rescue medication intakes due to measurement inaccuracies for bottle weights were considered as no intake.
Time Frame: From Day 1 up to Day 14 (End of Part 1)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: milligrams per kilogram per day
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1)
Number analyzed (Participants) | 24 | 45
milligrams per kilogram per day
  Average daily dose: number analyzed (Participants) | 24 | 44
  Average daily dose | 0.07 (0.154) | 0.46 (2.426)
  Modified average daily dose: number analyzed (Participants) | 24 | 44
  Modified average daily dose | 0.08 (0.160) | 0.11 (0.201)

7. Other Pre Specified Outcome: Serum Concentrations of Tapentadol (Part 1)
Description: Tapentadol serum concentrations were measured in participants in the tapentadol treatment arm (Part 1).
  All participants who had quantifiable serum concentrations during the Treatment Period were included in the descriptive pharmacokinetic analysis. Data from participants who vomited within 6 hours of administration of IMP during the Treatment Period were carefully assessed to decide if the data should be included in the pharmacokinetic analysis.
Time Frame: From Day 1 to Day 14 (End of Part 1)
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Groups:
- Tapentadol Prolonged-release (All Participants): The treatment group comprised 12 participants aged 6 years to less than 12 years and 33 participants aged 12 years to less than 18 years. Participants starting doses varied from 25 to 100 mg tapentadol PR twice daily depending on participant's weight. If necessary, doses were gradually increased up to a maximum dose defined per weight group.
  The highest dose defined for participants weighing 55 kg and more was 500 mg per day.
- Tapentadol Prolonged-release (6 Years to Less Than 12 Years): The treatment group comprised 12 participants aged 6 years to less than 12 years. Participants starting doses varied from 25 to 100 mg tapentadol PR twice daily depending on participant's weight. If necessary, doses were gradually increased up to a maximum dose defined per weight group.
  The highest dose defined for participants weighing 55 kg and more was 500 mg per day.
- Tapentadol Prolonged-release (12 Years to Less Than 18 Years): The treatment group comprised 33 participants aged 12 years to less than 18 years. Participants starting doses varied from 25 to 100 mg tapentadol PR twice daily depending on participant's weight. If necessary, doses were gradually increased up to a maximum dose defined per weight group.
  The highest dose defined for participants weighing 55 kg and more was 500 mg per day.
Arm/Group | Tapentadol Prolonged-release (All Participants) | Tapentadol Prolonged-release (6 Years to Less Than 12 Years) | Tapentadol Prolonged-release (12 Years to Less Than 18 Years)
Number analyzed (Participants) | 44 | 12 | 32
nanograms per milliliter
  Day 1: number analyzed (Participants) | 40 | 12 | 28
  Day 1 | 19.1 (19.57) | 17.2 (7.40) | 19.9 (22.99)
  Day 14: number analyzed (Participants) | 41 | 12 | 29
  Day 14 | 44.7 (34.17) | 35.6 (18.14) | 48.5 (38.59)

8. Other Pre Specified Outcome: Serum Concentrations of Tapentadol-O-glucuronide (Part 1)
Description: Tapentadol-O-glucuronide is a metabolite of tapentadol. The body transforms tapentadol into its metabolites so that it can be more easily/quickly removed from the body. Tapentadol-O-glucuronide serum concentrations were measured in participants who received tapentadol PR in Part 1.
  All participants who had quantifiable serum concentrations were included in the descriptive pharmacokinetic analysis. Data from participants who vomited within 6 hours of administration of IMP during Part 1 were carefully assessed to decide if they should be included in the pharmacokinetic analysis.
Time Frame: From Day 1 to Day 14 (End of Part1)
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Tapentadol Prolonged-release (All Participants) | Tapentadol Prolonged-release (6 Years to Less Than 12 Years) | Tapentadol Prolonged-release (12 Years to Less Than 18 Years)
Number analyzed (Participants) | 44 | 12 | 32
nanograms per milliliter
  Day 1: number analyzed (Participants) | 40 | 12 | 28
  Day 1 | 731.7 (840.02) | 603.2 (312.11) | 786.7 (984.42)
  Day 14: number analyzed (Participants) | 40 | 12 | 28
  Day 14 | 1557.3 (1187.24) | 1223.8 (511.27) | 1700.3 (1363.41)

9. Other Pre Specified Outcome: Palatability of Study Medication (Part 1, Day 8)
Description: Palatability was determined in Part 1 by asking the participant "How does the medication taste". The participant was requested to give a score on a 5-point hedonic faces rating scale in combination with a verbal rating. The response can range from really bad to really good.
Time Frame: Day 8 (Part 1)
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1)
Number analyzed (Participants) | 24 | 45
Participants
  Really bad | 0 | 0
  Bad | 0 | 2
  A bit bad/a bit good | 13 | 21
  Good | 7 | 12
  Really good | 3 | 6
  Missing | 1 | 4

10. Other Pre Specified Outcome: Palatability of Study Medication (Part 1, Day 14)
Description: as for outcome 9
Time Frame: Day 14 (Part 1)
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1)
Number analyzed (Participants) | 24 | 45
Participants
  Really bad | 0 | 0
  Bad | 0 | 1
  A bit bad/a bit good | 9 | 23
  Good | 9 | 11
  Really good | 6 | 9
  Missing | 0 | 1

11. Other Pre Specified Outcome: Acceptability of Study Medication (Part 1, Day 8)
Description: Acceptability of the study medication was determined in Part 1 by asking the participant "Swallowing the medication is...". The participant was requested to give a score on a 5-point hedonic faces rating scale in combination with a verbal rating. The response can range from really difficult to really easy.
Time Frame: Day 8 (Part 1)
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1)
Number analyzed (Participants) | 24 | 45
Participants
  Really difficult | 0 | 0
  Difficult | 0 | 3
  A bit difficult/a bit easy | 3 | 5
  Easy | 8 | 9
  Really easy | 12 | 24
  Missing | 1 | 4

12. Other Pre Specified Outcome: Acceptability of Study Medication (Part 1, Day 14)
Description: as for outcome 11
Time Frame: Day 14 (End of Part 1)
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1)
Number analyzed (Participants) | 24 | 45
Participants
  Really difficult | 1 | 1
  Difficult | 0 | 1
  A bit difficult/a bit easy | 2 | 7
  Easy | 8 | 16
  Really easy | 13 | 19
  Missing | 0 | 1

13. Other Pre Specified Outcome: Extent of Constipation (Part 2)
Description: Constipation was assessed using the modified constipation assessment scale (mCAS). This is an 8-item questionnaire where the observer has scored constipation on a nominal scale (no problem [score 0], some problem [score 1] or severe problem [score 2]). The response to an item could also be scored as "unable to assess".
  The Total Score can vary from 0-16; the higher the Total Score the higher the extent of constipation. A positive change from baseline to last assessment indicates a worsening, a negative change an improvement.
Time Frame: From baseline (Day 15 or switch) to last assessment (up to Day 379 of Part 2)
Population: Safety Set
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tapentadol in Part 2 After Tapentadol or Morphine in Part 1: Participants on tapentadol PR in Part 1 of the study continued on the current dose of tapentadol PR in Part 2 and if necessary could modify their tapentadol PR dosage. Participants who were randomized to morphine PR in Part 1 of the study were rotated to tapentadol PR in Part 2 with 70 percent of their current morphine equivalent dose or lower.The dosage could be increased gradually up to approximately 4.5 mg/kg body weight tapentadol PR twice daily.
  Tapentadol prolonged release
Arm/Group | Tapentadol in Part 2 After Tapentadol or Morphine in Part 1 | Observation Period After Tapentadol in Part 1 | Observation Period After Morphine in Part 1 | Observation Period After Tapentadol in Part 2
Number analyzed (Participants) | 36 | 18 | 14 | 26
units on a scale
  Baseline: number analyzed (Participants) | 35 | 17 | 14 | 25
  Baseline | 2.3 (2.4) | 1.8 (2.3) | 2.5 (2.5) | 1.5 (2.5)
  Last assessment: number analyzed (Participants) | 32 | 10 | 12 | 16
  Last assessment | 1.8 (2.7) | 0.4 (0.8) | 0.4 (1.2) | 0.8 (1.7)
  Change from baseline: number analyzed (Participants) | 32 | 9 | 12 | 15
  Change from baseline | -0.7 (3.3) | -1.4 (2.1) | -1.6 (1.7) | -1.4 (2.7)

14. Other Pre Specified Outcome: Change From Baseline in Subjective Opiate Withdrawal Scale (SOWS)
Description: Opiate withdrawal symptoms were assessed using the Subjective Opiate Withdrawal Scale (SOWS) questionnaire. The SOWS is designed to reflect common motoric, autonomic, musculoskeletal, and psychic signs and symptoms of opiate withdrawal. Each participant was requested to rate the first 15 items of the 16-item questionnaire for 7 days after last IMP intake. Participants rated the intensity of specific signs and symptoms on a scale of 0 (not at all) to 4 (extremely). The minimum overall score is 0, the maximum score is 64.
  SOWS Total Score at baseline (i.e., for Part 1 = Day 14-17, for Part 2 = Day 352-380, or the day after an early termination visit (Part 1/2)), and changes from baseline 2-7 days after last intake of IMP in Part 1 (= up to Day 23) and in Part 2 (= up to Day 386) are presented.
Time Frame: From Day 1 to Day 386 (End of Part 2 + 7 days)
Population: Safety Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 2)
Number analyzed (Participants) | 24 | 45 | 36
units on a scale
  Total score at baseline: number analyzed (Participants) | 9 | 9 | 23
  Total score at baseline | 4.0 (3.8) | 6.9 (7.6) | 6.1 (6.0)
  Change Day 2 after last IMP intake: number analyzed (Participants) | 10 | 10 | 25
  Change Day 2 after last IMP intake | -0.4 (2.0) | -1.7 (2.5) | -0.7 (2.8)
  Change Day 3 after last IMP intake: number analyzed (Participants) | 10 | 11 | 25
  Change Day 3 after last IMP intake | -1.6 (2.7) | -2.3 (4.9) | -0.3 (3.1)
  Change Day 4 after last IMP intake: number analyzed (Participants) | 10 | 12 | 27
  Change Day 4 after last IMP intake | -1.7 (4.4) | -3.9 (4.7) | -0.1 (3.6)
  Change Day 5 after last IMP intake: number analyzed (Participants) | 10 | 12 | 26
  Change Day 5 after last IMP intake | -1.6 (3.6) | -3.8 (5.1) | 0 (5.0)
  Change Day 6 after last IMP intake: number analyzed (Participants) | 9 | 12 | 25
  Change Day 6 after last IMP intake | -2.3 (3.6) | -3.6 (4.6) | -0.6 (3.1)
  Change Day 7 after last IMP intake: number analyzed (Participants) | 7 | 12 | 18
  Change Day 7 after last IMP intake | -2.7 (3.9) | -5.1 (6.3) | -1.4 (2.8)

15. Other Pre Specified Outcome: Time to Discontinuation (Lack of Efficacy) in Part 1
Description: The time to discontinuation from IMP due to lack of efficacy was planned to be analyzed for both treatment arms (tapentadol PR and morphine PR) in Part 1 of the trial. However, no participant was reported with early discontinuation from IMP due to lack of efficacy. Consequently, no time to discontinuation can be reported.
Time Frame: From first day in Part 1 (Day 1) to last day in Part 1
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Time to Discontinuation (Lack of Efficacy) in Part 2
Description: The time to discontinuation from IMP due to lack of efficacy was analyzed for tapentadol PR treatment in Part 2 of the trial.
Time Frame: From first day in Part 2 (Day 15) to last day in Part 2 (Day 379)
Population: Safety Set; 3 participants with early discontinuation from IMP due to lack of efficacy
Measure: Mean (Full Range); unit: weeks
Arm/Group | Tapentadol Prolonged-release (Part 2)
Number analyzed (Participants) | 3
weeks | 30.9 [9 to 36]

17. Other Pre Specified Outcome: Time to Discontinuation (Treatment Emergent Adverse Events) in Part 1
Description: The time to discontinuation from IMP due to treatment emergent adverse events (TEAEs) was analyzed for both treatment arms (tapentadol PR and morphine PR) in Part 1 of the study.
  Note that no participant discontinued due to a TEAE in the morphine PR arm, and 2 participants in the tapentadol PR arm.
Time Frame: From first day in Part 1 (Day 1) to last day in Part 1 (Day 14)
Measure: Mean (Full Range); unit: days
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1)
Number analyzed (Participants) | 24 | 45
days | NA [NA to NA] — No participant discontinued due to a TEAE in the morphine PR arm. | 3.0 [2 to 4]

18. Other Pre Specified Outcome: Time to Discontinuation (Treatment Emergent Adverse Events) in Part 2
Description: The time to discontinuation from IMP due to treatment emergent adverse events (TEAEs) was analyzed for tapentadol PR treatment in Part 2 of the study.
Time Frame: From first day in Part 2 (Day 15) to last day in Part 2 (Day 379)
Population: Safety Set; 3 participants discontinued due to treatment emergent adverse events.
Measure: Mean (Full Range); unit: weeks
Arm/Group | Tapentadol Prolonged-release (Part 2)
Number analyzed (Participants) | 36
weeks | 5.3 [3 to 24]

19. Other Pre Specified Outcome: Time to First Intake of Rescue Medication in the Open-label, Active-controlled Treatment Period (Part 1)
Description: Morphine oral solution could be given during Part 1 as rescue medication in both treatment groups. The dose per rescue medication intake was 1/6 of the total daily dose of the scheduled tapentadol or morphine PR intakes. Rescue medication administration times and doses were recorded.
  18 Participants in the morphine PR group and 27 participants in the tapentadol PR group had no documented intake of rescue medication between Day 1 and Day 14.
  Summary statistics were calculated based on participants with any intake, i.e., those that took at least 1 dose of rescue medication. The mean (standard deviation) time (hours) to first dose of rescue medication following the first dose of the IMP (on Day 1) is presented.
Time Frame: From Day 1 up to Day 14 (End of Part 1)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1)
Number analyzed (Participants) | 24 | 45
hours
  Participants with rescue medication intake: number analyzed (Participants) | 6 | 18
  Participants with rescue medication intake | 39.7 (63.75) | 74.6 (94.45)
  Participants with no rescue medication intake: number analyzed (Participants) | 18 | 27
  Participants with no rescue medication intake | NA (NA) — No documented intake of rescue medication between Day 1 and Day 14. | NA (NA) — No documented intake of rescue medication between Day 1 and Day 14.

ADVERSE EVENTS:
Time Frame: Adverse events were regularly assessed by the investigator using a standard set of questions. Treatment emergent adverse events (TEAEs) were collected from first dose (on Day 1) to last intake of IMP plus 72 hours (therapeutic reach).
Description: Part 1: TEAEs from first to last dose in Part 1 if participant continued on tapentadol PR in Part 2; from first to last dose in Part 1 + 72 hours (therapeutic reach) if participant did not continue on tapentadol PR in Part 2.
  Part 2: TEAEs from start of Part 2 to the last IMP intake in Part 2 + 72 hours (therapeutic reach).
Groups:
- Overall (Part 1): Overall (Part 1) includes all participants with a 2-week treatment with tapentadol PR or morphine PR tablets.
  One participant who completed the tapentadol PR treatment in Part 1 died in the Observation Period (Part 2; standard-of-care treatment, no IMP) due to progression of Ewing's sarcoma, which started progressing in Part 1. A second participant died in the Observation Period after Tapentadol in Part 1 due to serious progression of osteosarcoma with fatal outcome. The progression started in the Observation Period.
- Tapentadol Prolonged-release in Part 2: Tapentadol prolonged release in Part 2 comprises all participants who completed Part 1 (on tapentadol PR or morphine PR) and continued on or switched to an extended treatment with tapentadol PR for up to 12 months.
  No deaths were reported during treatment with tapentadol PR in Part 2. Following tapentadol PR treatment in Part 2, 1 participant died during the Observation Period (under standard-of-care treatment, no IMP) due to malignant neoplasm progression (sarcoma). The progression started in the Observation Period.
Arm/Group | Morphine Prolonged-release (Part 1) | Tapentadol Prolonged-release (Part 1) | Overall (Part 1) | Tapentadol Prolonged-release in Part 2
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/45 | 0/69 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/24 | 3/45 | 4/69 | 13/36
Other Adverse Events (participants affected / at risk) | 11/24 | 26/45 | 37/69 | 30/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine Prolonged-release (Part 1) (N=24) | Tapentadol Prolonged-release (Part 1) (N=45) | Overall (Part 1) (N=69) | Tapentadol Prolonged-release in Part 2 (N=36)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Breakthrough pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Movement disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dissociation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Limb operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine Prolonged-release (Part 1) (N=24) | Tapentadol Prolonged-release (Part 1) (N=45) | Overall (Part 1) (N=69) | Tapentadol Prolonged-release in Part 2 (N=36)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 6 (7) | 6 (7) | 3 (6)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4) | 7 (7) | 11 (11) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (5) | 10 (10) | 14 (15) | 11 (18)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Vomiting (Gastrointestinal disorders) | 7 (9) | 6 (6) | 14 (16) | 5 (5)
Fatigue (General disorders) | 3 (3) | 2 (2) | 5 (5) | 2 (3)
Pyrexia (General disorders) | 1 (1) | 3 (5) | 4 (6) | 2 (4)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 3 (3) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2) | 3 (9)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 4 (4) | 2 (2)
Dysarthria (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 6 (9) | 9 (12) | 10 (24)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any proposed presentation of the results of this trial before they are submitted for publication or public disclosure. Neither party (e.g., the sponsor, the coordinating investigator) has the right to prohibit publication or public disclosure unless it can be shown to affect possible patent rights.

DOCUMENTS (2):
  • Study Protocol (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT02151682/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT02151682/SAP_001.pdf